CLINICAL TRIAL: NCT07057258
Title: Injection Versus Suture Repair of Laryngeal Clefts, A Randomized, Controlled Trial
Brief Title: Injection Versus Suture Repair of Laryngeal Clefts
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Derek Lam, MD, MPH, Professor, American Academy of Otolaryngology-Head and Neck Surgery Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00027965
Record Dates: First submitted 2025-06-02; First posted 2025-07-09 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Laryngeal Cleft; Dysphagia
Keywords: endoscopic suture repair; injection laryngoplasty; pediatrics; otolaryngology; dysphagia; laryngeal cleft
MeSH Terms: conditions — Laryngeal cleft; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic suture repair (Experimental): Children receiving endoscopic suture repair of laryngeal cleft
  Interventions: Procedure: Endoscopic suture repair
- Injection laryngoplasty (Active Comparator): Children receiving injection of the interarytenoid space of laryngeal cleft
  Interventions: Procedure: Injection laryngoplasty

INTERVENTIONS:
Procedure: Endoscopic suture repair — Children receiving endoscopic suture repair of laryngeal cleft
  Arms: Endoscopic suture repair
Procedure: Injection laryngoplasty — Children receiving injection of the interarytenoid space for laryngeal cleft treatment
  Arms: Injection laryngoplasty

SUMMARY:
The purpose of the study is to learn more about a procedure that may be helpful for the participant's swallowing issues. The investigators are hoping to find out if one type of procedure is the same or better than another type of procedure at improving participant's issues with swallowing.

Participants will get one of two procedures. One is called injection laryngoplasty (IL) and injects a gel into the back wall of the participant's airway to prevent food and liquid from falling in. The other procedure is called endoscopic suture repair (ER) and uses sutures to sew together and build up the back wall of the participant's airway to prevent food and liquid from falling in. Participants will be asked to have a number of tests and procedures. These include a modified barium swallow study, in which the participant drinks and eats foods and liquids with barium in them and X-rays are used to assess how the food moves through the participant's body. This will be done before the procedure and 3 months after the procedure. The investigators will also give participants questionnaires to complete before and after the procedure.

DETAILED DESCRIPTION:
This study has 2 study groups.

* Group 1 will get IL for this condition.
* Group 2 will get ER for this condition

A computer will assign each participant to a group in no particular order. This is called randomization. Half of participants in this study will get IL. Half of participants will get ER. Each participant will have an equal chance of being in either group.

Neither the participants, the study doctor(s), nor the speech pathologist will know whether each participant will get the IL or ER. Only the surgeon will know which treatment the participant gets. The study is done this way because knowing which method the participant receives can change the results of the study.

If participants experience any serious side effects, the study doctor can find out which method they received so that any side effects can be treated properly.

Participants will need to have the following tests to find out if they can be in the study:

* Physical exam
* Demographic information/medical history
* Video fluoroscopic swallow study (VFSS) - X-ray videos that allow investigators to watch how food and liquids go down as a participant swallows them

If participant's screening tests show that they can take part in the study and they choose to be part of the study, they will also have to do the following tests:

* VFSS 3 months after the procedure
* Questionnaires asking about the emotional and physical burden of participant's swallowing issues, both before and after the procedure
* Overnight monitoring in the hospital after the procedure
* Follow up in clinic for up to 2 years after the procedure

Participant's medical records may be reviewed. Information reviewed may include treatment history, medications, surgeries, allergies, scans, and lab results.

Once participant's participation in the study ends, their medical provider(s) will help them choose the next step in their care.

ELIGIBILITY:
Inclusion Criteria:

* children aged 12 months - 10 years referred to a multi-disciplinary aerodigestive clinic with evidence of penetration or aspiration on VFSS, requiring any amount of thickening of liquids and unable to wean after 2-month trial of thickened liquids.

Exclusion Criteria:

* Cerebral palsy
* Down syndrome
* Prematurity < 28 weeks gestational age
* Hypoxic brain injury
* Any syndrome with significant hypotonia
* History of nothing by mouth (NPO) for > 1 month prior to assessment
* >50% of nutrition by G-tube
* Tracheostomy
* History of prior IL or ER

Ages: 12 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Resolution of penetration/aspiration | 3 months post operative
  No thickener needed on speech pathologist assessment of video fluoroscopic swallow study

SECONDARY OUTCOMES:
Compare change in recommended liquid thickness | at enrollment and 3 months post intervention
  The recommend liquid thickness according to speech pathologist assessment of video fluoroscopic swallow study review will be converted to a numerical scale and compared to pre-intervention recommended thickness to determine the degree of change after the intervention. The liquid thickness will be measured based on the IDDSI (International Dysphagia Diet Standardisation Initiative) Framework in which recommended liquid is scored as thin (0), slightly thick (1), mildly thick (2), moderately thick (3), or extremely thick (4). Higher scores indicate need for thicker liquids and therefore higher degree of dysphagia.
change in penetration/aspiration score | at enrollment and 3 months post intervention
  The score according to the Penetration-Aspiration scale rating of the video fluoroscopic swallow study data will be compared before and after the intervention. The Penetration-Aspiration scale includes: material does not enter the airway (1), material enters the airway, remains above the vocal folds, and is ejected from the airway (2), material enters the airway, remains above the vocal folds, and is not ejected from the airway (3), material enters the airway, contacts the vocal folds, and is ejected from the airway (4), material enters the airway, contacts the vocal folds, and is not ejected from the airway (5), material enters the airway, passes below the vocal folds, and is ejected into the larynx or out of the airway (6), material enters the airway, passes below the vocal folds, and is not ejected from the trachea despite effort (7), material enters the airway, passes below the vocal folds, and no effort is made to eject (8). Higher scores indicate higher degree of dysphagia.
change in feeding and swallowing impact survey (FSIS) scores | at enrollment and 3 months post intervention
  Survey data including FSIS will be analyzed and change in score will be calculated before and after the intervention. The FSIS is a validated survey that includes 18 statements that caregivers rate on a scale of 1 to 5 in which lower scores indicate better quality of life.
change in quality of life scores | at enrollment and 3 months post intervention
  Survey data including the Child Health Questionnaire (CHQ) for children aged five years and older or the Infant Toddler Quality of Life Questionnaire (ITQOL) for children aged under five years will be analyzed and change in score will be calculated before and after the intervention. The CHQ consists of 28 questions that assess the global quality of life of the child. The ITQOL consists of 47 questions that assess the global quality of life of the child. Based on the responses, the questionnaires are converted to a scale that ranges from 0 (worst possible score) to 100 (best possible score).
Change in laryngeal cleft quality of life (LC-QOL) scores | at enrollment and 3 months post intervention
  Survey data including LC-QOL will be analyzed and change in score will be calculated before and after the intervention. The LC-QOL is a 40 item questionnaire designed to assess quality of life in caregivers of patients with laryngeal cleft. Each item is scored from 0 to 5 in which lower scores indicate more significant negative impact on quality of life due to caring for a child with laryngeal cleft.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No